CLINICAL TRIAL: NCT00176722
Title: The Effect of Table Position on Intraocular Pressure (IOP) and Ocular Perfusion Pressure (OPP) During Prone Spine Surgery
Brief Title: Intraocular Pressure During Prone Spinal Surgery
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator is leaving the UMDNJ
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); New Jersey Eye Institute (Unknown)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120040320
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Spine Surgery; Vision Impairment
Keywords: Spine Surgery; Intraocular Pressure; lumbar or thoracic Spine Surgery in the prone position; and its association with visual change
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surgical: males & females undergoing spine surgery in the prone position
  Interventions: Other: table tilt

INTERVENTIONS:
Other: table tilt — One group randomized to table tilt. One group will be flat.

SUMMARY:
Postoperative visual loss resulting from surgical procedures not performed on the eye is a devastating outcome for the patient and poorly understood by the medical community. It is potentially a preventable complication. Diminished blood supply to the optic nerve, affecting both the anterior or posterior portions of the optic nerve, is the most common cause of postoperative visual loss. Other, less common causes include occlusion of the retinal artery and vein, a retinal embolism and cortical blindness. The incidence of postoperative visual loss increases in patients undergoing cardiopulmonary bypass and prone spinal surgery. Although the etiology of postoperative visual loss is unknown, it is thought to be multifactorial, and several potential risk factors have been identified, including degree of low blood pressure, preoperative hematocrit, external compression of the eye, amount of blood loss, prolonged duration of surgical time and lying in the face down position. The investigators believe this study is a unique opportunity to examine the mechanisms responsible for the antecedents to postoperative visual loss (POVL) and ischemic optic neuropathy (ION), a devastating complication of (usually) an elective surgical procedure. The purpose of this research is to try and determine the potential variables responsible for postoperative visual loss which will assist the medical community in devising methods for its prevention.

DETAILED DESCRIPTION:
Postoperative permanent visual loss is a rare but devastating complication of surgery estimated to occur after approximately 1/60,000 anesthetics. After procedures involving cardiopulmonary bypass and prone spinal surgery, the estimates are higher, 1/1600 to 1/1100, respectively and have led to the formation in July of 1999 of the Postoperative Visual Loss (POVL) Registry under the auspices of the American Society of Anesthesia (ASA) Committee on Professional Liability. The majority of reported cases as of early 2003 were associated with spine surgery (67%).

Of the spine cases, the majority were due to ischemic optic neuropathy (ION) (81%) followed by central retinal artery occlusion (13%) and unknown diagnosis (6%). Central retinal artery occlusion is characterized by periorbital edema, a cherry red spot at the fovea and monocular blindness. It is thought to be due to direct prolonged extraocular pressure on the globe and thus is preventable. Direct pressure on the eye is the etiology most often mentioned by spine surgeons in an attempt to explain all forms of postoperative visual loss.

Post anesthetic ION, affecting both the anterior and posterior portions of the optic nerve, however, is the more common diagnosis. The etiology is unclear but hypo perfusion of the optic nerve has been associated with multiple risk factors. The four patient factors are obesity, hypertension, diabetes and low preoperative hematocrit. There are five surgical factors, which include an operation of long duration, large blood loss, prone position, deliberate hypotension, and blood replacement strategies which increase the tissue fluid compartment while decreasing the hematocrit. ION occurs in patients who had their heads suspended in Mayfield tongs (18% of ION cases), virtually eliminating any source of external pressure. In addition, 58% of these patients had bilateral disease, making direct pressure less likely.

Thus, most POVL cases appear to be directly related to a change in retinal and/or optic nerve perfusion. The visual loss associated with anterior ION is caused by infarction in the watershed zones between the areas supplied by the posterior ciliary arteries, which are end arteries without anastomosis. Posterior optic neuropathy is thought to be caused by decreased oxygen delivery to the posterior portion of the optic nerve between the orbital apex and the entrance of the central retinal artery.

Critical to any discussion of perfusion to the eye is the concept of ocular perfusion pressure (OPP), defined as the difference between the mean arterial pressure (MAP) and the intraocular pressure (IOP). Unopposed decreases in MAP, increases in IOP or a combination of the two may result in hypo perfusion of the eye and can cause an ocular infarction at the level of the retina or optic nerve, leading to varying degrees of visual loss which is frequently bilateral and irreversible.

Animal data indicate that IOP increases with downward head tilting in the supine position, possibly due to increased episcleral venous pressure. Limited data for awake human volunteers indicate that IOP increases with supine positioning and is further elevated with head down tilting and prone positioning again possibly due to a rise in episcleral venous pressure.

This is a randomized prospective study examining the effect of the table position on intraocular pressure and ocular perfusion pressure during spine surgery.

Subjects will be recruited following the preoperative visit to the Neurosurgical office. An informed consent will be obtained after the consent for surgery is signed. A visual acuity exam will be performed with one of the study team members with the subject wearing corrective lenses on the morning of the surgery. The reactivity of the pupil will also be assessed via a penlight.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years of age who are mentally capable of providing an informed consent.
* Planned elective spinal surgery in which the modified Jackson table will be used.

Exclusion Criteria:

* Failure to provide an informed consent
* History of stroke
* Known history of corneal disease
* Known history of carotid disease
* Known history of sensitivity to cyclogyl and/or proparacaine HCL 0.5%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing spine surgery in the prone position.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-06; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
changes in intraocular pressure and retinal oximetry | over introperative time

CONTACTS AND LOCATIONS:
Overall Officials: Geordie Grant, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - University of Medicine & Dentistry - New Jersey Medical School, Newark, New Jersey
  - University of Medicine & Dentistry of NJ, Newark, New Jersey